CLINICAL TRIAL: NCT03263650
Title: Randomized Phase II Study of Olaparib Maintenance Following Cabazitaxel-Carboplatin Induction Chemotherapy in Men With Aggressive Variant Prostate Cancer (AVPC)
Brief Title: Study of Olaparib Maintenance Following Cabazitaxel-Carbo in Men With AVPC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: AstraZeneca (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0133; NCI-2018-01071 (Registry Identifier: NCI CTRP); 2017-0133 (Other: MD Anderson)
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer Aggressiveness; Prostate Carcinoma
Keywords: prostate cancer; genomic alterations; DNA damage repair; DDR pathway gene expression; aggressive-variant prostate carcinomas; small cell prostate carcinoma; neuroendocrine prostate carcinoma
MeSH Terms: conditions — Prostate Cancer, Hereditary, 7; Prostatic Neoplasms | interventions — cabazitaxel; Carboplatin; Prednisone; olaparib

STUDY DESIGN:
Intervention Model Description: All participants will receive 6 cycles of cabazitaxel and carboplatin before being randomized 2:1 to olaparib maintenance versus observation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cabazitaxel + Carboplatin (Experimental): Cabazitaxel, Cabazitaxel and Carboplatin intravenously on day 1 of cycles 1-6. Prednisone by mouth twice daily on days 1-21 of cycles 1-6.
  Interventions: Drug: Cabazitaxel; Drug: Carboplatin; Drug: Prednisone 5Mg
- Olaparib Maintenance (Experimental): Participants randomized to receive Olaparib by mouth twice daily on Day 1 of cycle 7.
  Interventions: Drug: Olaparib
- Observation Only (No Intervention): Participants randomized to observation only beginning cycle 7.

INTERVENTIONS:
Drug: Cabazitaxel — 25mg/m2 administered intravenously over 60 minutes on day 1 of cycles 1-6; given before carboplatin.
  Other Names: Jevtana
  Arms: Cabazitaxel + Carboplatin
Drug: Carboplatin — AUC 4 administered intravenously over 60 minutes on day 1 of cycles 1-6
  Other Names: Paraplatin
  Arms: Cabazitaxel + Carboplatin
Drug: Prednisone 5Mg — 5 mg administered by mouth twice daily on days 1-21 of cycles 1-6.
  Arms: Cabazitaxel + Carboplatin
Drug: Olaparib — Administered by mouth twice daily at a dose of 300 mg by mouth twice daily, dispensed on Day 1 of cycle 7 to participants randomized to receive olaparib maintenance and every 21 days thereafter until the participant completes the study, withdraws from the study or the closure of the study.
  Other Names: Olaparib Pill
  Arms: Olaparib Maintenance

SUMMARY:
The goal of this clinical research study is to learn if olaparib, when given after treatment with cabazitaxel, carboplatin, and prednisone, can help to control aggressive variant prostate cancer (AVPC). The safety of these drugs will also be studied.

This is an investigational study. Cabazitaxel and carboplatin are FDA approved and commercially available for the treatment of certain types of prostate cancer. Prednisone is FDA-approved and commercially available as a corticosteroid. Olaparib is FDA approved and commercially available for the treatment of certain types of ovarian cancer. The combination of cabazitaxel and carboplatin followed by olaparib in this study is investigational.

The study doctor can describe how the study drugs are designed to work.

Up to 96 participants will be enrolled on this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in a roll of dice) to 1 of 2 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group. You will have a 2 in 3 chance of being assigned to Group 1 and a 1 in 3 chance of being assigned to Group 2:

* If you are in Group 1, you will receive olaparib.
* If you are in Group 2, you will not receive olaparib.

All participants will receive cabazitaxel and carboplatin.

You and the study staff will know to which group you have been assigned.

Study Drug Administration:

Each study cycle is 21 days.

You will receive cabazitaxel by vein over 60 minutes on Day 1 of Cycles 1-6. You will then receive carboplatin by vein over 60 minutes on Day 1 of Cycles 1-6.

You will take 1 tablet of prednisone by mouth 2 times each day of Cycles 1-6.

You will be given standard drugs to help decrease the risk of side effects (for example, filgrastim) before and/or after each dose of cabazitaxel and continuing through several days. Your doctor will describe these drugs to you in more detail, including how they are given and any side effects you may expect.

If you are in Group 1, you will take tablets of olaparib 2 times by mouth each day starting on Day 1 of Cycle 7. Swallow the whole tablet or tablets. Do not chew, crush, divide, or dissolve the tablets. If you vomit shortly after taking your olaparib tablet you can retake a new dose as long as you can see that the tablet came out whole. You should take the doses at the same time each day (or within 2 hours of the scheduled times). Do not take the dose if you forget and it is more than 2 hours since your scheduled time. Take olaparib at least 1 hour after and 2 hours before eating.

If you are in Group 2, you will receive standard of care treatment and follow-up after Cycle 6. The study doctor will tell you more about what this may mean for you.

Length of Treatment:

You will receive carboplatin and cabazitaxel for up to 6 cycles. If you are in Group 1, you may continue receiving olaparib for as long as the doctor thinks it is in your best interest. You may no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

Study Visits:

On Day 1 of Cycles 1-6:

* You will have a physical exam.
* Blood (up to 5 tablespoons) will be drawn for routine tests, biomarker testing, tumor marker testing, and to measure your PSA level. At some of these visits, this sample will also be used for CTC testing. You must fast for up to 12 hours before the Cycle 4 visit.
* Urine will be collected for tumor marker testing.
* At Cycle 4 only, you will have a bone scan and either MRIs or CT scans to check the status of the disease.

After Cycle 6, you will have a second tumor biopsy for biomarker testing to compare to the one taken at screening. The type of biopsy you have will depend on where the disease has spread and/or what the doctor thinks is in your best interest. The doctor will discuss with you the type of biopsy you will have.

On Day 1 of Cycle 7:

* Blood (up to 5 tablespoons) will be drawn to check your testosterone levels, biomarker testing, and for tumor marker testing.
* You will have an EKG.
* You will have a bone scan and either MRIs or CT scans.

On Day 1 of Cycles 8-10:

* You will have a physical exam.
* Blood (up to 5 tablespoons) will be drawn for routine tests, tumor marker testing, biomarker testing, and to measure your PSA level. At some of these visits, this sample will also be used for CTC testing.
* Urine will be collected for tumor marker testing.

After Cycle 10, you will only have study visits every 3 cycles. Beginning on Day 1 of Cycle 13, every 3 cycles (Cycles 13, 16, 19, and so on):

* You will have a physical exam.
* Blood (up to 5 tablespoons) will be drawn for routine tests, tumor marker testing, biomarker testing, and to measure your PSA level. At some of these visits, this sample will also be used for CTC testing. You must fast for up to 12 hours before the visits at Cycle 10 and every 3 cycles after that.
* Urine will be collected for tumor marker testing.
* You will have a bone scan and either MRIs or CT scans to check the status of the disease.
* You will have an EKG.

If you have severe side effects, you may return to the clinic more often so the study doctor can check on your health.

End of Study Visit:

When you leave the study, the following tests and procedures will be performed:

* You will have a physical exam.
* You will have a bone scan and either MRIs or CT scans to check the status of the disease.
* You will have an EKG.
* Blood (about 3 tablespoons) will be drawn for routine tests, tumor marker testing, and to measure your PSA level. You must fast for up to 12 hours before this visit.
* Urine will be collected for tumor marker testing.

Follow-Up:

About every 6 months after the end-of-study visit, the study staff will check your health. This will be done either by a chart review or a phone call. If you are called, this call will last about 5 minutes. These calls will stop if you withdraw from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Provision of informed consent for genetic research. If a patient declines to participate in the genetic research, there will be no penalty or loss of benefit to the patient. The patient will not be excluded from other aspects of the study described in this Clinical Study Protocol, so long as they consent to that part.
3. Patients must agree to tissue collection for correlative studies at the specified timepoints. If patient has undergone a recent tissue collection without intervening treatment since, that can be retrieved and is deemed of sufficient quantity by the PI to undertake the proposed correlative studies, it may be used as the baseline.
4. Male aged 18 years and above.
5. Histologically or cytologically confirmed prostate carcinoma.
6. Presence of metastatic disease documented on imaging studies (bone scan, computed tomography (CT) and/or magnetic resonance imaging (MRI) scans).
7. Patients must meet at least one of the following AVPC criteria: i. Histologically proven small cell (neuroendocrine) prostate carcinoma ii. Exclusive visceral metastases. iii. Predominantly lytic bone metastases identified by plain x-ray or CT scan. iv. Bulky (>/= 5cm in longest dimension) lymphadenopathy or high-grade tumor mass in prostate/pelvis. v. Low PSA (</= 10ng/mL) at initial presentation (prior to androgen ablation or at symptomatic progression in the castrate-setting) plus high volume (>/= 20) bone metastases. vi. Elevated serum lactate dehydrogenase (>/=2 x upper limit of normal) or elevated serumcarcinoembryonic antigen (>/= 2 x upper limit of normal ) in the absence of other etiologies. vii. Short interval (</= 180 days) to castrate-resistant progression following initiation of hormonal therapy. viii. Known loss or mutation (by CLIIA certified molecular testing, IHC and/or DNA sequencing) in at least 2 of the following: Tp53, RB1 and PTEN.
8. (continued from Inclusion Criteria #7: viiii. Patients who have castration -resistant disease progression per RECIST but do not meet PCWG3 PSA progression criteria
9. Patients must have documented evidence of progressive disease as defined by any of the following: a) PSA progression: minimum of 2 rising values (3 measurements) obtained a minimum of 7 days apart with the last result being at least >/= 1.0 ng/mL; b) New or increasing non-bone disease (RECIST); c) Positive bone scan with 2 or more new lesions (PCWG3). d) Increasing symptoms unequivocally attributed to disease progression as judged by the treating physician and the PI.
10. Surgically or ongoing medically castrated, with baseline testosterone levels of </= 50 ng/dL </= 2.0 nM).
11. Eastern Cooperative Oncology Group (ECOG) Performance Status of </=2.
12. Patients must have normal organ and bone marrow function measured within 7 days prior to administration of study treatment as defined below: i. Hemoglobin >/= 10.0 g/dL dL (unless due to bone marrow infiltration by tumor, in which case hemoglobin >/=8gdL is allowed). Patient may have blood transfusions prior to study enrollment. ii. Absolute neutrophil count (ANC) >/= 1.5 x 10^9/L (unless due to bone marrow infiltration by tumor, in which case ANC >1,000/mm3 is allowed) iii. White blood cells (WBC) >3x10^9/L (unless due to bone marrow infiltration by tumor, in which case WBC >2x109/L is allowed) iv. No features suggestive of myelodysplastic syndrome/acute myeloid leukemia on peripheral blood smear v. Platelet count >/= 100 x 10^9/L (unless due to bone marrow infiltration by tumor, in which case platelet >/=50,000/ mm3 is allowed) vi. Total bilirubin </=1.5 x institutional upper limit of normal (ULN) (except for patients with known Gilbert's disease).
13. (continued from Inclusion Criteria #11 vii. aspartate aminotransferase (serum glutamine oxaloacetic transminase) and alanine aminotransferase (serum glutamic pyruvic transaminase) </= 2.5 x institutional upper limit of normal (unless liver metastases are present in which case it must be </= 5x ULN) viii. Calculated creatinine clearance (Cockcroft-Gault Equation) >/= 40 mL/min.
14. Able to swallow study drugs whole as a tablet/capsule.
15. Patients who have partners of childbearing potential (e.g. female that has not been surgically sterilized or who are not amenorrheic for >/= 12 months) must be willing to use a method of birth control in addition to adequate barrier protection as determined to be acceptable by the investigator during the study and for 13 weeks after last study drug administration. Please note that the efficacy of hormonal contraception may be decreased if administered with olaparib.
16. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at MD Anderson)
2. Previous enrolment or randomization in the present study
3. Any prior treatment for castration-resistant prostate cancer (CRPC) with carboplatin, cisplatin, cabazitaxel or olaparib.
4. Patients whose disease is refractory (defined as evidence of disease progression while on drug or within 3 months of its discontinuation) to more than 2 lines of chemotherapy given for CRPC. Any number of chemotherapies to which the patient's disease is not refractory are allowed, as long as time on treatment did not exceed 6 months (counted from day 1 of cycle 1 to day 1 of the last cycle of treatment).
5. Patients who have not recovered from adverse events secondary to systemic therapy (except for luteinizing hormone-releasing (LHRH) hormone agonist or antagonist treatment for prostate cancer, and bisphosphonates or receptor activator of Nf kappa (RANK) ligand inhibitors for bone strengthening), major surgery or radiotherapy for the treatment of prostate cancer to a grade </= 2.
6. Persistent toxicities (>/= common terminology criteria for adverse events grade 2) with the exception of alopecia, caused by previous cancer therapy.
7. Chronic use of known strong CYP3A4 inhibitors (e.g. ketoconazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin, voriconazole, nefazodone, posaconazole, ritonavir, lopinavir/ritonavir, indinavir, saquinavir, boceprevir, telaprevir and nelfinavir), moderate CYP3A4 inhibitors (e.g. amprenavir, aprepitant, atazanavir, ciprofloxacin, crizotinib, darunavir/ritonavir, diltiazem, erythromycin, fluconazole, fosamprenavir, imatinib, verapamil), strong CYP3A4 inducers (e.g. phenytoin, rifampicin, carbamazepine, St.John's Wort, phenobarbital) and moderate CYP3A4 inducers (e.g. bosentan, efavirenz, etravirine, modafinil and nafcillin). Concomitant use of these drugs with olaparib is not allowed. Patients may undergo limited courses of them prior to starting olaparib but will be required to have >/= 5 week washout period from phenobarbital, and >/=3 week washout period from the rest, before randomization.
8. Active uncontrolled infection ( patients completing a course of antibiotic or antiviral therapy whose infection is deemed to be controlled may be allowed on study after discussion with the PI; the PI will serve as the final arbiter regarding eligibility).
9. Active or symptomatic viral hepatitis or chronic liver disease.
10. A diagnosis or suspicion of myelodysplastic syndrome/acute myeloid leukemia.
11. A history of pneumonitis or extensive bilateral lung disease of non-malignant etiology.
12. A malignancy [other than the one treated in this study] which required radiotherapy or systemic treatment within the past 5 years, or has a >/= 30% probability of recurrence within 24 months (except for adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the Ta urothelial carcinomas).
13. Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, superior vena cava syndrome, extensive bilateral lung disease on high-resolution computed tomography scan, uncontrolled seizures or any psychiatric disorder that prohibits obtaining informed consent.
14. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
15. Patients with symptomatic uncontrolled brain metastases or spinal cord compressions. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 28 days prior to treatment.
16. Patients with a known hypersensitivity to the olaparib, carboplatin or cabazitaxel.
17. Prisoners or subjects who are involuntarily incarcerated.
18. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer study: Histologically or cytologically confirmed prostate carcinoma.
Enrollment: 96 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) of men with AVPC treated with 6 cycles of cabazitaxel + carboplatin followed by olaparib maintenance versus observation | Up to one year from time of randomization
  Progression Free Survival (PFS) calculated as the time from randomization until any one of the following events occurs, whichever comes first:
  * Documented disease progression
  * Start of a new therapy in the absence of progression
  * Death in the absence of progression

SECONDARY OUTCOMES:
Genomic alterations in DNA damage repair (DDR) pathway genes induced and/or selected by carboplatin and cabazitaxel chemotherapy [biopsy #2 vs biopsy #1]: Association with clinical outcome (PFS>6 months) | Up to one year
Rate of adverse events possibly, probably or definitely attributable to olaparib following cabazitaxel plus carboplatin in men with AVPC | Up to one year
Overall survival (OS) of men with AVPC treated with 6 cycles of cabazitaxel + carboplatin followed by olaparib maintenance vs observation | Up to one year
Response evaluation criteria in solid tumors (RECIST) and prostate specific antigen (PSA) response rate (RR) to cabazitaxel + carboplatin induction, and to olaparib maintenance in men with AVPC | Up to one year
Association between DDR pathway gene expression changes following carboplatin + cabazitaxel chemotherapy and clinical outcome (PFS>6 months) | Up to one year
Collection and archiving of serum, plasma, and urine samples in study patients for later hypothesis generating associations | Up to one year

CONTACTS AND LOCATIONS:
Overall Officials: Ana M. Aparicio, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org